CLINICAL TRIAL: NCT01167686
Title: Phase 2 Study of Gardemont S.A Food Supplement on Symptoms of Upper Respiratory Illness
Brief Title: Effects of Gardemont S.A Food Supplement on Upper Respiratory Illness
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Collaborators: Ben-Gurion University of the Negev (Other); Clalit Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: k008/2010
Record Dates: First submitted 2010-07-21; First posted 2010-07-22 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Respiratory Infections
Keywords: Respiratory infection; Viral infection; Food supplement; Goldtrain Plus (GT+)
MeSH Terms: conditions — Respiratory Tract Infections; Virus Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Food supplement (Experimental): Half of the subjects participating in the trial (91) will recieve four tablets of the food supplement (Gardemont Goldrain Plus) three times a day for seven consecutive days from inclusion.
  Interventions: Dietary Supplement: Gardemont Goldtrain Plus (GT+)

INTERVENTIONS:
Dietary Supplement: Gardemont Goldtrain Plus (GT+) — Four tablets of 760 mg of GT+ administered three times a day for seven consecutive days and similar placebo tablets given to the control arm

SUMMARY:
General:Prospective, randomized, double blind controlled trial of the food supplement GOLDTRAIN PLUS, to assess its safety and efficacy in comparison to placebo in subjects with upper respiratory infection.

Hypothesis: The food supplement GOLDTRAIN PLUS will be superior to placebo in shortening the time to recovery from the disease symptoms.

Study design and outcome measures:Study population of 182 generally healthy subjects with acute respiratory infection randomized in 1:1 ratio to active supplement versus placebo treatment, with randomization stratified by site. The study supplement administration will be continued for 7 days, and patient global assessment (PGA) will be the main primary measurement tool, based on a self-reporting questionnaire filled and monitored every 12 hours for 7 consecutive days. Throat and nasal swabs determining type of viral infection, will be taken at inclusion of patient and a number of blood tests at the end of treatment to look for any adverse effects of the medication.

Analysis and conclusion: All data-from the filled questionnaires, clinical follow up and laboratory studies will be analyzed by multivariate analysis to determine the efficacy of the supplement and its correlation to the clinical and laboratory parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent
2. Age eligible (18 ≤ Age ≤ 90)
3. Respiratory infection with or without fever-

Exclusion Criteria:

1. Evidence of the bacterial infection
2. Symptoms suggestive of other than respiratory system illness (i.e. diarrhea, abdominal pain, skin rash, urinary symptoms).
3. Hospitalisation is planned
4. Surgery within previous 2 months
5. Pregnancy (women at childbirth age should have a urine beta-HCG test performed)
6. Subject with known renal dysfunction (creatinine ≥ 2 mg/dL)
7. Subject has history of debilitating liver dysfunction with elevation of liver enzymes and bilirubin levels to ≥ ULN
8. Participation in the active follow-up phase of another clinical study of an investigational drug or device
9. Known hypercalcemia -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-11 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Patient Global Assessment (PGA) | Seven days
  Patient global assessment (PGA) will be a primary measurement, based on the self-reporting answer to the following question: "What is your overall feeling as compared to the first day of treatment: worse, same or better". Time from the enrollment to the first 12 hours when the subject reports on a sustained improvement in symptoms (two consequent 12 hours periods) will be a primary outcome. The study supplement administration will be continued for 7 days.

SECONDARY OUTCOMES:
Rate of safety composite | 30 days
  Death, hospitalizations, serious adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Zvi Bentwich, MD, Study Director — Ben-Gurion University of the Negev
Locations (1):
- Revivim and Mashabei Sadeh Clalit Clinics, Beersheba, Israel